CLINICAL TRIAL: NCT04923022
Title: The Effect of Therapeutic Exercise and Vegan Diet on Pain and Quality of Life in Young Women With Chronic Idiopathic Neck Pain.
Brief Title: Therapeutic Exercise and Vegan Diet on Pain and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Mustafa Savaş Torlak, Principal Investigator, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41901325-050.99
Record Dates: First submitted 2021-06-02; First posted 2021-06-11 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Chronic Idiopathic Neck Pain
MeSH Terms: interventions — Diet, Vegan; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vegan diet (Experimental): Participants with chronic neck pain who will be on a vegan diet will follow a diet program prepared by an expert dietitian under the supervision of an endocrinologist. In this diet program, a diet that includes grains, fruits, vegetables, legumes, as well as dairy products and eggs, known as lacto-ovo vegetarian, will be applied. Consumption of meat, poultry, fish, seafood and processed food and beverages will not be allowed. There will be no calorie restriction in the diet, and the diet will be arranged according to the amount of calories calculated by the expert dietitian according to BMI. The diet will last for eight weeks. Individuals who follow a diet will be constantly checked by the workers with the mobile device application (My Fitness Pal®).
  Interventions: Other: Vegan Diet
- Therapeutic exercise (Experimental): The participants in the therapeutic exercise group will perform the following therapeutic exercises for eight weeks, 3 days a week, accompanied by a specialist physiotherapist.
  1. The patient, sitting in the cervical spine neutral position, performs flexion, extension and rotation of the cervical spine, unloaded and in the maximum possible range of motion.
  2. While the patient is in the supine position, she performs passive lateral mobilization to the neck with the help of a physiotherapist.
  3. In the supine position, the patient performs isometric neck flexion, lateral flexion and rotation movements against the manual resistance given by the physiotherapist
  4. The patient lying on his back does isometric neck extension movement against gravity
  5. The patient performs isometric neck flexion, lateral flexion and rotation movements against the elastic band in the sitting position
  Interventions: Other: Therapeutic exercise
- Control group (No Intervention): Participants in this group will not receive any intervention.

INTERVENTIONS:
Other: Vegan Diet — Participants with chronic neck pain who will be on a vegan diet will follow a diet program prepared by an expert dietitian under the supervision of an endocrinologist. In this diet program, a diet that includes grains, fruits, vegetables, legumes, as well as dairy products and eggs, known as lacto-ovo vegetarian, will be applied. Consumption of meat, poultry, fish, seafood and processed food and beverages will not be allowed. There will be no calorie restriction in the diet, and the diet will be arranged according to the amount of calories calculated by the expert dietitian according to BMI. The diet will last eight weeks. Individuals who follow a diet will be constantly checked by the workers with the mobile device application (My Fitness Pal®).
  Arms: Vegan diet
Other: Therapeutic exercise — Individuals in the therapeutic exercise group will perform therapeutic exercises for eight weeks, 3 days a week, accompanied by a specialist physiotherapist.
  Arms: Therapeutic exercise

SUMMARY:
45 sedentary volunteer female individuals whose age range is between 18-25 years and diagnosed with chronic idiopathic neck pain by a specialist physical therapy doctor will participate in the study. Participants will be randomly divided into three groups: vegan diet group (n=15), therapeutic exercise group (n=15) and control group (n=15). Participants with chronic neck pain who will be on a vegan diet will follow a diet program prepared by an expert dietitian under the supervision of an endocrinologist. In this diet program, a diet that includes grains, fruits, vegetables, legumes, as well as dairy products and eggs, known as lacto-ovo vegetarian, will be applied. Consumption of meat, poultry, fish, seafood and processed food and beverages will not be allowed. There will be no calorie restriction in the diet, and the diet will be arranged according to the amount of calories calculated by the expert dietitian according to BMI. The diet will last eight weeks. Individuals who follow a diet will be constantly checked by the workers with the mobile device application (My Fitness Pal®). Individuals in the therapeutic exercise group will perform therapeutic exercises for eight weeks, 3 days a week, accompanied by a specialist physiotherapist.The aim of this study is to compare the Effect of Therapeutic Exercise and Vegan Diet on Pain and Quality of Life in Young Women with Chronic Idiopathic Neck Pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-25,
* neck pain for at least 3 months,
* VAS score greater than 5

Exclusion Criteria:

* using regular analgesic,
* having had neck surgery,
* the presence of neurological or specific problems in the neck (vertebral fracture, inflammation, infection, etc.),
* cortisone use,
* pregnancy,
* serious chronic diseases,
* those with serious psychiatric disorders
* Individuals who received physical therapy within 3 months
* Antidepressant use

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 1 minute
  Body mass index will be calculated as weight/height2
Visual Analog Scale (VAS) | 2 minutes
  Pain intensity was evaluated with the Visual Analogue Scale (VAS). The VAS consists of a 10 cm long horizontal line. 0 means "no pain " and 10 means "unbearable severe pain". Individuals marked the level of corresponding to pain they felt on the 10 cm line, and the values of the marked places were calculated with a 100-millimeter ruler
Neck Disability Index (NDI) | 10 minutes
  This index consists of 10 parts and the each part of index has 6 different answers. In these 10 parts, there are answers about the severity of neck pain, personal care of the individual, lifting, reading, headache, concentration, work life, driving, sleep and leisure activities. It is scored as 0 (no pain and functional limitation) and 5 (the most severe pain and maximum limitation). In the NDI, 0-4 points were stated as no disability, 5-14 points mild disability, 15-24 points moderate disability, 25-34 points severe disability and 35 points above complete disability
Short Form 36 | 15 minutes
  this questionnaire consists of 36 questions covering eight domains of health and wellbeing corresponding subscales, whichare used to estimate a physical (PCS) and a mental com-ponent score (MCS).The sub-parameters of the test are physical function, physical role difficulty, emotional role difficulty, energy, mental health, social functionality, pain and general health perception. A minimum of 0 and a maximum of 100 points can be obtained from the test. A high scores from the test indicates well-being.
Tampa Scale of Kinesiophobia (TSK-17) | 15 minutes
  The kinesiophobia was evaluated using the Tampa Scale of Kinesiophobia (TSK-17). The validity and reliability of the scale was performed by Yılmaz et al.
  There is a 4-point likert scoring in the scale. The total score ranges between 17 and 68. A high value on the TSK-17 indicates a high degree of kinesiophobia and a cut-off score was developed by Vlaeyen et al., where a score of 37 or over is considered a high score.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)